CLINICAL TRIAL: NCT06327308
Title: Evaluation of Cirrhotic Cardiomyopathy by Cardiac MRI in Patients Waiting for Liver Transplant. A Multicenter Prospective Pilot Study. (CARDIO-FIBROCIR)
Brief Title: Evaluation of Cirrhotic Cardiomyopathy by Cardiac MRI in Patients Waiting for Liver Transplant.
Acronym: CARDIOFIBROCIR
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/803
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2023-09

CONDITIONS: Cirrhosis
Keywords: Cirrhosis; cirrhotic cardiomyopathy; Liver Transplantation; MRI
MeSH Terms: conditions — Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with cirrhosis requiring liver transplantation
  Interventions: Diagnostic Test: MRI; Biological: Blood sampling

INTERVENTIONS:
Diagnostic Test: MRI — The examination lasts between 45 minutes and one hour. The patient lies down in the MRI tube. He is fitted with headphones that muffle the noise produced by the machine and enable him to receive instructions from the technician. Four electrodes are applied to his chest to continuously record his heartbeat. Finally, his chest is covered with a plastic plate, which receives the MRI signals needed to form the image. Acquiring an MRI image takes between 2 and 20 seconds. To ensure that image quality is not impaired by respiratory movements, images are acquired in apnea. The technician will ask the patient to hold his or her breath repeatedly throughout the examination.
Biological: Blood sampling — Additional blood will be drawn for dosing acylcarnitines, copeptin, interleukin-6 (IL-6), LPS-Binding Protein (LBP), Phospholipid TransferProtein (PLTP)/Cholesteryl Ester Tranfer Protein (CETP) activity, and for plasma banking. The volume of blood will be 20 ml in total (5 ml for each assay) at each visit. Patients participating in this study will have 3 visits. Total blood volume will therefore be 20 x 3, or 60 ml for the 3 visits.

SUMMARY:
The aim of this multicenter prospective observational pilot study is to describe the evolution of myocardial fibrosis in cirrhotic patients before and after liver transplantation (LT). Through multimodal analysis of myocardial function and architecture, and analysis of specific markers of inflammation, we aim to explore the following hypotheses: 1) systemic inflammation promotes myocardial fibrosis in cirrhotic patients and could be an early marker of cirrhotic cardiomyopathy; 2) LT allows resolution of myocardial fibrosis by preventing the bacterial translocation that favors the development of deleterious systemic inflammation.

DETAILED DESCRIPTION:
Cirrhotic patients with an indication for LT and undergoing pre-transplant assessment will be eligible for this study. All included patients will undergo myocardial Magnetic Resonance Imaging (MRI) at the time of inclusion, then at a second visit that will be planned as close as possible to the expected date of LT or at 9 months in the absence of LT, then 12 months after LT or 21 months after inclusion for non-transplanted patients. Markers of systemic inflammation will be analyzed at these same time points.

* Primary outcome : to describe the evolution of the percentage of myocardial fibrosis on cardiac MRI before and 12 months after LT in cirrhotic patients.
* Secondary outcomes

  1. To describe the evolution of the percentage of myocardial fibrosis at 9 months and 21 months in non-transplanted patients.
  2. To estimate the prevalence of cirrhotic cardiomyopathy in cirrhotic patients before and 12 months after LT.
  3. To describe the relationship between plasma 3-hydroxymyristate (3-HM) concentration and the level of myocardial fibrosis estimated by myocardial extracellular volume (MECV) before and 12 months after LT
  4. To describe the relationship between several markers of inflammation (CRP, procalcitonin, copeptin, IL-6) or proteins modulating the degree of inflammation (LPS-binding protein (LPB), Phospholipid Transfer Protein (PLTP), Cholesteryl Ester Transfer Protein (CETP)) and the level of myocardial fibrosis estimated by MECV, before and 12 months after LT.
  5. To describe, in liver transplanted patients, the evolution of the percentage of myocardial fibrosis before and 12 months after LT according to the degree of immunosuppression.
  6. To describe, in liver transplanted patients, the occurrence of cardiovascular events according to the cirrhotic cardiomyopathy status, from inclusion (i.e., placement on the transplant waiting list) to transplantation.
  7. To describe the occurrence of cardiovascular events according to the cirrhotic cardiomyopathy status in the 12 months following LT.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion of cirrhotic patients when registering on the liver transplant list
* Women who have been menopausal for at least 24 months, surgically sterilized, or, for women of childbearing age, use an effective method of contraception (oral contraceptives, contraceptive injections, intrauterine devices, double-barrier method, contraceptive patches)
* Signature of an informed consent form indicating that the subject has understood the purpose and procedures required by the study and that he or she agrees to participate in the study and to comply with the requirements and restrictions inherent in the study
* Patient with a social security system or beneficiary of such a system.

Exclusion Criteria:

* Minor or over 70 years old
* Transplant Patient
* Patient with a TIPS
* Known cardiorespiratory disease including portopulmonary hypertension and coronary artery disease
* Uncontrolled hypertension with interventricular septal thickness ≥ 15 mm
* Hemodynamic instability
* Type 1 diabetes
* Current bacterial infection
* HIV infection (or unknown HIV status)
* Contraindications for MRI including pacemaker, implantable defibrillators, electrosystolic pacing probe, Swan-Ganz probe, postoperative epicardial electrodes, Starr-Ewards metal ball valves, insulin pumps, ferromagnetic vascular clips, ocular and otological implants, ocular ferromagnetic foreign bodies, renal failure with a GFR < 30 mL/min/1.73 m², contraindication to contrast media, patient unable to maintain apnea for a few seconds, claustrophobia
* Inability to receive informed information in patients with severe encephalopathy who do not have a trusted person
* Refusal to agree to participation by signing the information and consent form as defined
* Patient under guardianship, curatorship, Legal incapacity or limited legal capacity
* Patient deprived of liberty
* Pregnant woman or breastfeeding
* Subject unlikely to cooperate in the study and/or low cooperation anticipated by the investigator
* Subject without health insurance
* Subject being in the period of exclusion from another study or provided for by the "national volunteer file"

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with cirrhosis requiring LT and eligible for LT according to a pre-liver transplant assessment that does not contraindicate LT. Patients listed for fulminant hepatitis or early re-transplantation will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure | sixth month-21th month after inclusion
  Difference in myocardial extracellular volume (MECV) on cardiac MRI between the pre-LT visit (visit 2) and 12 months after LT (visit 3). If patients are transplanted less than 6 months after the inclusion visit, visit 2 will not be performed and the reference visit will be visit 1.

SECONDARY OUTCOMES:
Prevalence of cirrhotic cardiomyopathy according to 2019 criteria [Izzy M, et al. Hepatology 2020;71:334-45], echocardiographic signs of left ventricular systolic and diastolic dysfunction : | 33 months
  * Systolic dysfunction: left ventricular ejection fraction ≤ 50% and/or absolute value of left ventricular global longitudinal strain value < 18%.
  * Diastolic dysfunction if ≥ 3 criteria among the following:
    * Mitral e' wave velocity < 7 cm/s ;
    * Mitral e' wave / E wave ratio ≥ 15 ;
    * Indexed left atrial volume > 34 mL/m² ;
    * Tricuspid regurgitation velocity > 2.8 m/s.
Analysis of the association between myocardial extracellular volume (MECV) (explained variable) and plasma 3-HM concentration (explanatory variable). | 33 months
  The concentration of 3-hydroxy-myristate will be in pg/ml. Analysis of the association between myocardial extracellular volume (MECV) (explained variable) and plasma 3-HM concentration (explanatory variable) will be based on the observation of the point cloud.
Analysis of the association between myocardial extracellular volume (MECV) and the concentration of markers of inflammation (CRP, procalcitonin, copeptin, IL-6) and proteins modulating the degree of inflammation (LBP, PLTP, CETP). | 33 months
  Analysis of the association between myocardial extracellular volume (MECV) and the concentration of markers of inflammation (CRP, procalcitonin, copeptin, IL-6) and proteins modulating the degree of inflammation (LBP, PLTP, CETP) will be based on the observation of the point cloud.
Analysis of the association between the difference in MECV in transplant recipients between visit 2 and visit 3 according to the degree of immunosuppression, measured by mean residual tacrolemia in the 12 months post-LT. | sixth month-21th month after inclusion
Number, type and cumulative incidence of cardiovascular events (heart failure, rhythm disorders, etc.) according to cirrhotic cardiomyopathy status occurring between inclusion and LT. | 33 months
Number, type and cumulative incidence of cardiovascular events (heart failure, rhythm disorders, etc.) occurring between inclusion and LT, according to cirrhotic cardiomyopathy status. | 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Thierry THEVENOT, MD, PHD, Study Director — Centre Hospitalier Universitaire de Besancon; Delphine WEIL, MD, Principal Investigator — Centre Hospitalier Universitaire de Besancon; Camille BESCH, MD, Principal Investigator — CHU Strasbourg; Mouni BENSENANE -OUSSALAH, MD, Principal Investigator — CHRU Nancy; Marianne LATOURNERIE, MD, Principal Investigator — CHU Dijon
Locations (4):
- France (4):
  - CHU Besancon - Hopital Minjoz, Besançon
  - CHU Dijon - Hopital François Mitterrand, Dijon
  - CHRU Nancy - Hôpital de Brabois, Nancy
  - CHU Strasbourg - Hopital de HautePierre, Strasbourg